CLINICAL TRIAL: NCT03756207
Title: Clinical Study on Efficacy and Safety of Multidisciplinary Bladder-preservation Therapy for Muscle-invasive Bladder Cancer in China
Brief Title: Multidisciplinary Bladder-preservation Therapy for Bladder Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2018183
Record Dates: First submitted 2018-11-15; First posted 2018-11-28 (Actual); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Bladder Cancer
Keywords: multidisciplinary; bladder cancer; bladder-preservation
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: In this study, the investigators plan to prospectively recruit 80 muscle-invasive bladder cancer patients, who don't want to receive radical cystectomy or are not candidates for radical cystectomy, treated with multidisciplinary bladder-preservation therapy from Nov 2018 to Dec 2020 in Peking University Third Hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multidisciplinary Therapy (Experimental): Multidisciplinary bladder-preservation therapy: Maximal transurethral resection followed by radiotherapy with concomitant radio-sensitizing chemotherapy
  Interventions: Procedure: multidisciplinary bladder-preservation therapy

INTERVENTIONS:
Procedure: multidisciplinary bladder-preservation therapy — Maximal transurethral resection followed by radiotherapy with concomitant radio-sensitizing chemotherapy

SUMMARY:
A multidisciplinary approach has led to the development of bladder-preservation therapy using maximal transurethral resection followed by radiotherapy with concomitant radio-sensitizing chemotherapy for muscle-invasive bladder cancer.

DETAILED DESCRIPTION:
Multidisciplinary management improves complex treatment decision making in cancer care, but its impact for bladder cancer has not been documented. Although radical cystectomy (RC) has long been the standard of care for the management of muscle-invasive bladder cancer (MIBC), a multidisciplinary approach has led to the development of bladder-preservation therapy using maximal transurethral resection (TURBt) followed by radiotherapy with concomitant radio-sensitizing chemotherapy for MIBC. There are no randomized-controlled data comparing radical cystectomy with multidisciplinary bladder-preservation therapy (MBPT) available for comparison. However, observational data continues to support the use of MBPT as an acceptable alternative for patients with MIBC who wish to preserve their bladder or are not candidates for cystectomy because it may result in equivalent disease outcomes in select patients and offers the benefit of maintaining a functioning urinary system with subsequent improvements in quality of life. But there are also lots of issues need to be studied, such as the patient selection, approaches for completeness of TURBt, choices of radio-sensitizing chemotherapy, accuracy of radiotherapy and so on. In this study, the investigators plan to prospectively recruit 80 MIBC patients, who don't want to receive RC or are not candidates for RC, treated with MBPT from Nov 2018 to Dec 2020 in Peking University Third Hospital. The investigators will collect, compare and analyze their clinic-pathological data before and after MBPT, in order to confirm the safety and efficacy of MBPT for MIBC in China. At the same time, the investigators want to find out the patients who are not suitable for MBPT and the approach which can improve the efficacy of MBPT, as a result, the investigators intend to make a standard MBPT approach for Chinese MIBC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Bladder urothelial carcinoma
2. Clinical stage: T2-T4, non-metastasis
3. Eastern Cooperative Oncology Group score (ECOG)≤ 1, Karnofsky performance score≥ 70
4. Patients don't want to receive RC or are not candidates for RC
5. Normal bladder function

Exclusion Criteria:

1. History of abdominal and pelvic radiotherapy
2. History of other malignant tumor
3. Pregnant or lactating patients
4. Severe comorbidity: cardiac infarction, arrhythmia, heart failure, et al

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Complete response rate | 6-8 weeks after chemoradiation
  Response to MBPT depending on cystoscopy, TURBt, or urinary cytology
Disease specific survival (DSS) time | From date of treatment initiation until the date of death due to bladder cancer, assessed up to 60 months.
  Events were defined as death attributable to bladder cancer. The time to DSS was the interval between treatment initiation and death due to bladder cancer, or the most recent follow-up if no event occurred.
Overall survival (OS) time | From date of treatment initiation until the date of death due to any cause, assessed up to 60 months.
  Events were defined as death due to any cause. The time to OS was the interval between treatment initiation and death, or the most recent follow-up if no event occurred.

SECONDARY OUTCOMES:
Quality of life score 1 | 6-8 weeks after chemoradiation
  Assessed by EORTC Quality of life questionaire (QLQ)-30
Quality of life score 2 | 6-8 weeks after chemoradiation
  Assessed by EORTC QLQ-Bladder Cancer 30

CONTACTS AND LOCATIONS:
Overall Officials: Yi Huang, MD, Principal Investigator — Department of Urology, Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China